CLINICAL TRIAL: NCT00437190
Title: Pivotal IDE Study of the BRYAN(R) Cervical Disc Prosthesis in the Treatment of Degenerative Disc Disease
Brief Title: Pivotal IDE Study of the BRYAN(R) Cervical Disc Prosthesis in the Treatment of DDD Versus ACDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRYAN(R) Cervical Disc IDE
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Radiculopathy; Myelopathy; Cervical Degenerative Disc Disease
Keywords: Cervical Disc Replacement; Spondylotic radiculopathy; Spondylotic myelopathy; Myelopathy; Radiculopathy
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases | interventions — Transplantation, Homologous; Bone Plates; Total Disc Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterior Cervical Discectomy Fusion (Active Comparator)
  Interventions: Device: ATLANTIS™ Cervical Plate System and allograft
- BRYAN Cervical Disc Prosthesis (Experimental): BRYAN Cervical Disc Prosthesis is a cervical intervertebral disc prosthesis designed to provide for motion like the normal cervical functional spinal unit.
  Interventions: Device: BRYAN Cervical Disc Prosthesis

INTERVENTIONS:
Device: ATLANTIS™ Cervical Plate System and allograft — Control treatment is commercially available allograft (without bone matrix paste) used in conjunction with the Medtronic Safamor Danek ATLANTIS™ Cervical Plate System.
  Other Names: cervical plate; plate; fusion; cervical fusion
  Arms: Anterior Cervical Discectomy Fusion
Device: BRYAN Cervical Disc Prosthesis — The intent is to treat stable degenerative disc disease by implanting the BRYAN Cervical Disc Prosthesis to provide motion like the normal cervical functional spinal unit.
  Other Names: disc; cervical disc; artificial disc; BRYAN
  Arms: BRYAN Cervical Disc Prosthesis

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of the BRYAN(R) Cervical Disc Prosthesis in treating single-level degenerative disc disease of the cervical spine.

DETAILED DESCRIPTION:
Bryan(R) Cervical Disc Prosthesis is indicated in skeletally mature patients for reconstruction of the disc from C3 to C7 following single level discectomy for intractable radiculopathy and/or myelopathy.

ELIGIBILITY:
Inclusion Criteria:

The indication studied was degenerative disc disease (DDD) at a single level between C3 and C7 for any combination of disc herniation with radiculopathy, spondylotic radiculopathy, disc herniation with myelopathy, or spondylotic myelopathy.

The following additional inclusion criteria had to be present:

* At least 6 weeks unsuccessful conservative treatment, except in cases of myelopathy requiring immediate treatment (e.g., acute onset of clinically significant signs);
* Requirement for surgical treatment demonstrated by CT, myelography and CT, and/or MRI;
* Skeletally mature (≥ 21 years of age);
* Preoperative Neck Disability Index score of ≥ 30 and at least one clinical sign associated with level to be treated;
* Willing to sign informed consent and comply with protocol.

Exclusion Criteria:

Subjects were excluded if they had any of the following:

* Any of the following at the treated level:

  * Significant cervical anatomical deformity; e.g., ankylosing spondylitis, rheumatoid arthritis, etc.
  * Moderate to advanced spondylosis. Patients who demonstrate advanced degenerative changes. Such advanced changes are characterized by any one or combination of the following: bridging osteophytes, marked reduction or absence of motion, collapse of the intervertebral disc space of greater than 50% of its normal height;
  * Radiographic signs of subluxation greater than 3.5 mm;
  * Angulation of the disc space more than 11 degrees greater than adjacent segments;
  * Significant kyphotic deformity or significant reversal of lordosis;
* Axial neck pain as the solitary symptom;
* Previous cervical spine surgery;
* Metabolic bone disease, such as osteoporosis, defined as a BMD T-score equal to or worse than 2.5. If significant radiolucence is detected, a BMD scan in the spine, wrist, and femoral neck must be obtained.
* Active systemic infection or infection at the operative site;
* Known allergy or to titanium, polyurethane, or ethylene oxide residuals;
* Concomitant conditions requiring steroid treatment;
* Diabetes mellitus requiring daily insulin management;
* Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index;
* A medical condition that may interfere with the postoperative management program, such as advanced emphysema or Alzheimer's disease;
* A medical condition that may result in patient death prior to study completion: unstable cardiac disease, active malignancy;
* Pregnant;
* Current or recent alcohol and/or drug abuser requiring intervention;
* Signs of being geographically unstable, such as recent or pending divorce, or high level of job dissatisfaction.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2003-06; Primary Completion 2006-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Improvement in patient pain and ability to function | 24 months
  The self-administered Neck Disability Index patient questionnaire is used to assess patient pain and ability to function. A successful outcome will be declared if: Postoperative Score - Postoperative Score is ≥ 15.

CONTACTS AND LOCATIONS:
Overall Officials: Rick C Sasso, MD, Principal Investigator — Indiana Spine Group
Locations (38):
- United States (38):
  - Barrow Neurosurgical Associates, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Silicon Valley Spine Institute, Campbell, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Bay Area Spine Institute, Walnut Creek, California
  - North Florida Regional Medical Center, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Emory Orthopedics and Spine Center, Atlanta, Georgia
  - Northwestern University Department of Neurosurgery, Chicago, Illinois
  - University of Chicago Hospitals Section of Neurosurgery, Chicago, Illinois
  - Chicago Inst. of Neurosurgery and Neuro Research, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Indiana Spine Group, Indianapolis, Indiana
  - Neurosurgery Associates, Scarborough, Maine
  - Maryland Brain & Spine, Annapolis, Maryland
  - Neurosurgery of Kalamazoo, Kalamazoo, Michigan
  - Marquette General Brain & Spine Center, Marquette, Michigan
  - Cervical Spine Specialists, Edina, Minnesota
  - Twin Cities Spine Center, Minneapolis, Minnesota
  - Columbia Orthopaedic Group, Columbia, Missouri
  - Washington University Orthopedics, St Louis, Missouri
  - Spine Nevada, Reno, Nevada
  - Rochester Brain and Spine Neuro, Rochester, New York
  - Upstate Orthopedics, Syracuse, New York
  - Crouse Hospital, Syracuse, New York
  - Carolina Neurosurgery and Spine Specialists, Charlotte, North Carolina
  - Wake Forest University School of Medicine - Dept. of Neurosurgery Medical Center, Winston-Salem, North Carolina
  - Neurosurgical Network, Inc., Toledo, Ohio
  - Kellogg MD Brain & Spine, Portland, Oregon
  - Oregon Neurosurgery, Springfield, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Southeastern Spine Institute, Mt. Pleasant, South Carolina
  - Neurosurgical Associates, Nashville, Tennessee
  - NeuroSpine Consultants, PA, Plano, Texas
  - Neurosurgery Associates, Salt Lake City, Utah
  - University of Wisconsin Medical School, Madison, Wisconsin

REFERENCES:
- [Background] Sasso RC, Anderson PA, Riew KD, Heller JG. Results of cervical arthroplasty compared with anterior discectomy and fusion: four-year clinical outcomes in a prospective, randomized controlled trial. J Bone Joint Surg Am. 2011 Sep 21;93(18):1684-92. doi: 10.2106/JBJS.J.00476. PMID 21938372
- [Background] Heller JG, Sasso RC, Papadopoulos SM, Anderson PA, Fessler RG, Hacker RJ, Coric D, Cauthen JC, Riew DK. Comparison of BRYAN cervical disc arthroplasty with anterior cervical decompression and fusion: clinical and radiographic results of a randomized, controlled, clinical trial. Spine (Phila Pa 1976). 2009 Jan 15;34(2):101-7. doi: 10.1097/BRS.0b013e31818ee263. PMID 19112337
- [Derived] Arnold PM, Anderson KK, Selim A, Dryer RF, Kenneth Burkus J. Heterotopic ossification following single-level anterior cervical discectomy and fusion: results from the prospective, multicenter, historically controlled trial comparing allograft to an optimized dose of rhBMP-2. J Neurosurg Spine. 2016 Sep;25(3):292-302. doi: 10.3171/2016.1.SPINE15798. Epub 2016 Apr 29. PMID 27129045